CLINICAL TRIAL: NCT04632966
Title: A Prospective, Open-Label, Dose-Escalation Phase 1 Study of Intra-Articular Administration of an Allogeneic Human Placental Tissue Particulate (PTP-001) for the Treatment of Knee Osteoarthritis
Brief Title: Safety Study of PTP-001 for Treating Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KOA-20-01
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Open-label, dose-escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTP-001 - Low Dose (100 mg) (Experimental): intra-articular injection of 100 mg PTP-001 resuspended with 4 mL of normal saline
  Interventions: Biological: Biological: PTP-001
- PTP-001 - High Dose (200 mg) (Experimental): intra-articular injection of 200 mg PTP-001 resuspended with 4 mL of normal saline
  Interventions: Biological: Biological: PTP-001

INTERVENTIONS:
Biological: Biological: PTP-001 — allogeneic placental tissue particulate

SUMMARY:
Evaluation of safety, tolerability, and efficacy of a single intra-articular (IA) injection of PTP-001, an allogeneic placental tissue particulate, in individuals with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This open-label, dose-escalation study is expected to enroll 20 participants, 40-80 years of age and test two doses (low and high dose) of PTP-001, an allogeneic placental tissue particulate, in two unique cohorts of 10 participants each. Each participant will receive a single intra-articular (IA) injection of PTP-001. Following the completion of the first cohort in which 10 participants (Kellgren-Lawrence Grade 2 or 3 knee OA) will be treated with the low dose of PTP-001, safety data will be reviewed by an independent Data and Safety Monitoring Board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Male or female, aged 40 to 80 years
* Symptomatic knee OA with Kellgren-Lawrence radiographic classification of 2 or 3
* Non-responsive after at least 3 months of conservative therapy for knee OA
* Females of childbearing potential must have negative pregnancy test result prior to treatment and must commit to highly effective methods of contraception for at least 6 months after treatment
* Willingness to report oral analgesic treatment used for knee pain and to discontinue analgesic treatment for knee pain in 24 hours prior to each study visit
* Willingness to limit use of pain rescue medication to oral acetaminophen for management of painful knee OA flare

Exclusion Criteria:

* Body mass index (BMI) ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 with condition that warrants weight loss surgery
* Presence of active infection of index knee or systemic infection requiring treatment within 3 months of Screening
* Administration of IA injection within 3 months of Screening
* Significant acute injury to index knee within 3 months of Screening
* Surgery to index knee within 6 months of Screening or planned surgery to index knee within 6 months after Screening
* Unstable index knee joint
* History of radiation therapy of index knee
* Known vascular or neurological disorder affecting the index knee
* Osteonecrosis of either knee
* Clinical diagnosis of inflammatory arthritis
* Clinical diagnosis of autoimmune disease affecting the musculoskeletal system
* Use of any other investigational therapy within 3 months of Screening or planned for the duration of the study
* Current anti-coagulant use
* History of receiving a solid organ or hematologic transplant
* History of malignancy or radiotherapy within 5 years of Screening, except for basal or squamous cell carcinoma of the skin
* Use of immunosuppressive or chemotherapeutic agents within 5 years of Screening
* Known allergy to local anesthetics or allograft tissues
* Known history of hepatitis
* Known history of thrombotic or thromboembolic phenomena.
* Known history of primary or secondary immunodeficiency disorders
* Presence of concurrent medical condition that, in the investigator's judgement, could compromise participant safety or interfere with the required study assessments and study participation.

Note: Other protocol defined inclusion/exclusion criteria apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of local and systemic treatment emergent adverse events (AEs) and incidence of abnormal laboratory and immunogenicity panels | Baseline to Week 52
  Incidence of local and systemic treatment emergent adverse events (AEs), including clinical laboratory and immunogenicity panels, after a single intra-articular injection of PTP-001.

SECONDARY OUTCOMES:
Western Ontario and McMaster University (WOMAC) Pain Responder Rate | Week 26 and Week 52
WOMAC Physical Function Responder Rate | Week 26 and Week 52
Change from baseline in pain of the index knee, by evaluating the WOMAC Pain subscale score (the possible total score ranging from 0-50 for pain) | Baseline to Week 52
  WOMAC Numerical Rating Scale (NRS) 3.1 questionnaire is a health status measure questionnaire of 24 questions comprising 3 subscales (pain, stiffness and physical function). WOMAC A (measure of pain) is measured on 11-point NRS ranging from 0 (none) to 10 (extreme), where higher score represents higher pain.
Change from baseline in physical function of the index knee, by evaluating the WOMAC Physical Function subscale score (the possible total score ranging from 0-170 for Physical Function) | Baseline to Week 52
  WOMAC Numerical Rating Scale (NRS) 3.1 questionnaire is a health status measure questionnaire of 24 questions comprising 3 subscales (pain, stiffness and physical function). WOMAC C (measure of physical function) is measured on 11-point NRS ranging from 0 (none) to 10 (extreme), where higher score represents higher pain.
Change from baseline in patient global assessment of OA, by assessing the participants assessment of how they are doing considering arthritis in index knee (the possible answers include "Very Good", "Good", "Acceptable", "Poor", "Very Poor" | Baseline to Week 52
Change from baseline in health-related quality of life, by assessing the items from the Short Form 36 (SF-36) survey | Baseline to Week 52
  The SF-36 measures 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health (the possible total normalized score ranges from 0-100). Higher scores on the SF-36 indicate better health status.

OTHER OUTCOMES:
Change from baseline in biochemical markers (CTX-II & PRO-C2) | Baseline to Week 52
  * Urinary CTX-II samples
  * Serum PRO-C2 samples
Change from baseline in joint space width of the index knee, assessed radiographically (OARSI radiographic scoring) | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Annunziato Amendola, MD, Principal Investigator — James R. Urbaniak, MD, Duke Sports Science Institute
Locations (2):
- United States (2):
  - James R. Urbaniak, MD, Duke Sports Science Institute, Durham, North Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flannery CR, Seaman SA, Buddin KE, et al. Characterization and preclinical efficacy of PTP-001, a novel human tissue biologic in development for the treatment of OA. Osteoarthritis Cartilage. 2020 Apr;28(Supplement 1):S487-S489. doi: 10.1016/j.joca.2020.02.763
- [Background] Flannery CR, Seaman SA, Buddin KE, Nasert MA, Semler EJ, Kelley KL, Long M, Favret J, Pavesio A, Loeser RF. A novel placental tissue biologic, PTP-001, inhibits inflammatory and catabolic responses in vitro and prevents pain and cartilage degeneration in a rat model of osteoarthritis. Osteoarthritis Cartilage. 2021 Aug;29(8):1203-1212. doi: 10.1016/j.joca.2021.03.022. Epub 2021 May 20. PMID 34023528